CLINICAL TRIAL: NCT02545491
Title: Implementation of Care for Child Development and Implications on Early Childhood Development: A Pilot Study in Lebanon
Brief Title: Implementation and Adoption of Care for Child Development in Day Care Centers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: American University of Beirut Medical Center (Other)
Collaborators: World Vision (Other); Ministry of Public Health, Lebanon (Unknown)
Responsible Party: Principal Investigator, Lama Charafeddine, Assistant Professor in Clinical Pediatrics, MD FAAP, American University of Beirut Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: PED.DS.03
Record Dates: First submitted 2015-08-25; First posted 2015-09-10 (Estimated); Last update posted 2018-07-06 (Actual); Status verified 2018-07

CONDITIONS: Child Development
Keywords: CCD; Child development; daycare; caregiver
MeSH Terms: interventions — Child Development

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Care for Child Development group (Experimental): Training of caregivers on the Care for Child Development (CCD) program, in addition to the training on Infant and Young Child feeding program by World Vision.
  Interventions: Behavioral: Care for Child Development (CCD) program; Behavioral: Infant and Young Child feeding training by World Vision
- World Vision Lebanon training group (Active Comparator): caregivers will receive training in Infant and Young Child Feeding (WV-IYCF) offered by World Vision.
  Interventions: Behavioral: Infant and Young Child feeding training by World Vision

INTERVENTIONS:
Behavioral: Care for Child Development (CCD) program — The Care for Child Development (CCD) Program developed by World Health Organization (WHO) /UNICEF provides recommendations for stimulating child development through play and communication activities.
  Arms: Care for Child Development group
Behavioral: Infant and Young Child feeding training by World Vision — Training on breastfeeding benefits, solid introduction and food safety

SUMMARY:
Background: Responsive stimulation and/or enhanced nutrition interventions delivered to children through health programs shows improved cognitive, language, and motor, and the social-emotional status. This could benefit young children in Lebanon and worldwide to improve their developmental potential.

Aim: This study aims to implement Care for Child Development (CCD) intervention for children aged 0-3 years within a supportive environment in Day Care Centers and to investigate its effectiveness on early child development.

Methodology: CCD program will be implemented in 10 randomly selected daycare centers in Lebanon where three providers in each center will be trained (CCD-group). Another group of 10 day care centers will serve as controls (WV-group). 228 Children in each group will receive either early stimulation based on CCD and education from the World Vision Infant and Young Child Feeding (WV-IYCF) project (CCD-group) or education from the WV-IYCF project (WV-group). Caregivers' knowledge and behaviors will be assessed before and after the intervention using a predetermined questionnaire and behavioral checklist. Early child development will be assessed using Ages and Stages Questionnaire-3 (ASQ-3) and Bayley Scale for infant Development (BSID-III).

Expected Outcome: Implementation of CCD program in day care centers will be feasible and will lead to enhanced early child development. This study will serve as a prototype for program implementation throughout the country and the region.

DETAILED DESCRIPTION:
This study aims at testing the implementation and effectiveness of the CCD program on early child development in selected day care centers in Beirut. It is being conducted in collaboration with World Vision and the Lebanese Ministry of Public Health.

Day Care centers are invited by the ministry of health to participate in this proposed study.

After securing the approval of the Center's director, caregivers working at those day care centers are being invited to participate in this study.

Those caregivers who agree to participate will receive either training on the CCD program AND early child nutrition from World Vision (Infant & Young Child Feeding Project WV-IYCFP) (Intervention group) or training on early child nutrition from WV-IYCFP only (control group).

The Care for Child Development (CCD) Program developed by World Health Organization (WHO) /UNICEF provides caregivers with recommendations for stimulating child development through play and communication activities.

WV-IYCFP provides activities related to raising awareness on breastfeeding and complementary food introduction to optimize child nutrition.

The Intervention group (CCD-Group) consists of 10 day care centers chosen randomly. Three caregivers from each center (total 30 caregivers) will attend a day-and-a-half CCD training at the Center of Excellence for Early Child Development at AUBMC. In addition, they will participate in the World Vision activities related to the Infant & Young Child Feeding Project (WV-IYCFP). The day care centers in this group will receive a manual including early child development concepts and techniques to be used as a reference.

The Control group (WV-Group) consists of 10 day care centers chosen randomly. Three caregivers from each center (total 30 caregivers) will participate in activities related to the WV-IYCFP.

Caregivers in both groups will be asked to take a knowledge assessment questionnaire on child development before and after each training, then at 6months and 12 months after the intervention.

In both groups, caregivers' behavior in early child stimulation will be assessed before and after the trainings. Caregivers will be observed delivering child care as per each center's routine; their behavior will be assessed using a predetermined behavioral check list developed based on the CCD program.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 0 to 3 years registered in the selected daycare centers.

Exclusion Criteria:

* Children diagnosed with medical conditions that might affect developmental assessment, or who are older than the specified ages will not be included in the study.

Max Age: 3 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 136 (Actual)
Dates: Start 2015-01; Primary Completion 2017-11 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
Enhancing child development. (developmental scores by BSID-III ) | one year
  Children in the CCD-group will have better developmental scores by BSID-III compared to those in the WV- group.

SECONDARY OUTCOMES:
Caregivers' knowledge (measured by pre and post assessement test) | one year
  Caregivers in the intervention group will have at least 25% improvement in the 12 items knowledge assessment questionnaire after the intervention.
Caregivers' behavior (measured by behavioral observation using predetermined checklist) | one year
  Caregivers' behavioral checklist scores (after the intervention) will be of at least 8 out of 10 for those in the intervention group.

CONTACTS AND LOCATIONS:
Overall Officials: Durriyah Sinno, MD, Principal Investigator — American University of Beirut Medical Center
Locations (1):
- American University of Beirut, Beirut, Lebanon

REFERENCES:
- [Background] Anderson LM, Shinn C, Fullilove MT, Scrimshaw SC, Fielding JE, Normand J, Carande-Kulis VG; Task Force on Community Preventive Services. The effectiveness of early childhood development programs. A systematic review. Am J Prev Med. 2003 Apr;24(3 Suppl):32-46. doi: 10.1016/s0749-3797(02)00655-4. PMID 12668197
- [Background] Bryanton J, Beck CT. Postnatal parental education for optimizing infant general health and parent-infant relationships. Cochrane Database Syst Rev. 2010 Jan 20;(1):CD004068. doi: 10.1002/14651858.CD004068.pub3. PMID 20091558